CLINICAL TRIAL: NCT02368483
Title: The Effectiveness of Neuromuscular Training of the Lower Limb Muscles in Reducing the Hip Symptoms in Patients With Symptomatic Femoroacetabular Impingement: a Prospective Intervention Study
Brief Title: Conservative Treatment in Patients With Symptomatic Femoroacetabular Impingement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Responsible Party: Principal Investigator, Nicola Maffiuletti, PhD, Schulthess Klinik
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAI conservative treatment 1
Record Dates: First submitted 2015-01-29; First posted 2015-02-23 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Symptomatic Femoroacetabular Impingement

ARMS (1):
- Neuromuscular training (Experimental)
  Interventions: Other: Neuromuscular training

INTERVENTIONS:
Other: Neuromuscular training — Neuromuscular training for the hip and lower limb muscles.The training program is divided into 3 phases, and includes specific exercises for improving the hip range of motion, muscle strength of the hip and lower limb muscles, as well as the trunk stability and coordination. The intervention lasts 12 weeks. Patients will train 2 times/week with a physical therapist and 2 times/weeks alone at home.

SUMMARY:
This is a single-group, prospective, intervention study. A total of 30 participants with unilateral symptomatic femoroacetabular impingement will be included into the study. The intervention consists in neuromuscular training for the lower limb muscles (12 weeks, 2 times/week supervised training, 2 times/week home training). The training includes physical exercises routinely used worldwide in clinical settings. No control intervention group was included into the study because nowadays there is no standard conservative treatment for patients with symptomatic femoroacetabular impingement. Assessments will be performed at (1) baseline, (2) mid-intervention, (3) end-intervention, and (4) follow-up. Clinical, functional, neuromuscular and self-reported parameters will be collected during assessments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral symptomatic FAI according to clinical, radiographic and magnetic resonance imaging criteria
* Living place: Canton of Zurich or neighbouring Cantons
* Signed written informed consent to participate into the study

Exclusion Criteria:

* Previous hip surgery
* Any surgery to the lower limbs in the prior 6 months
* Congenital/developmental dysplasia
* Hip osteoarthritis
* Initiation of opioid analgesia and corticosteroid injection for hip pain within the prior 30 days
* BMI >35 kg/m2
* Significant cardiorespiratory diseases

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Hip Function as measured using the Hip Outcome Score questionnaire | Change from Baseline in Hip Function at 12 weeks
  Hip Function was assessed using the Hip Outcome Score. The Hip Outcome score is a questionnaire used to evaluate hip function during daily and sport activities. Two independent scores are obtained: one for activities of daily living and one for sport activities.

SECONDARY OUTCOMES:
Hip Muscle Strength as measured using dynamometry | Change from Baseline in Hip Muscle Strength at 12 weeks
  Hip abduction, adduction, internal rotation and external rotation isometric maximal voluntary contraction strength is evaluated with hand-held dynamometry. Hip flexion and extension isometric maximal voluntary contraction strength is evaluated with isokinetic dynamometry.
Movement Control Quality as measured using a visual rating scale | Change from Baseline in Movement Control Quality at 12 weeks
  Overall body movement pattern quality is visually assessed during the performance of 5 lower extremity functional tests (single-leg squat, lunge, hop lunge, single-leg bridge, single-leg ventral plank).

CONTACTS AND LOCATIONS:
Locations (1):
- Schulthess Clinic, Zurich, Switzerland

REFERENCES:
- [Derived] Casartelli NC, Bizzini M, Maffiuletti NA, Sutter R, Pfirrmann CW, Leunig M, Naal FD. Exercise Therapy for the Management of Femoroacetabular Impingement Syndrome: Preliminary Results of Clinical Responsiveness. Arthritis Care Res (Hoboken). 2019 Aug;71(8):1074-1083. doi: 10.1002/acr.23728. Epub 2019 Jul 9. PMID 30133164